CLINICAL TRIAL: NCT00076401
Title: Phase II Trial of Motexafin Gadolinium (MGd) in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Study of Motexafin Gadolinium for the Treatment of Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0216
Record Dates: First submitted 2004-01-21; First posted 2004-01-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Leukemia; Leukemia, Lymphocytic, Chronic
Keywords: CLL; chronic lymphocytic leukemia; relapsed chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; Leukemia; Motexafin gadolinium; Chronic leukemia; Lymphocytic leukemia, chronic
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin gadolinium

SUMMARY:
The purpose of this study is to determine if the drug motexafin gadolinium will be an effective treatment for patients who have chronic lymphocytic leukemia (CLL) that has come back after treatment or that has stopped responding to treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Refractory or relapsed CLL
* ECOG performance status score of 0, 1, or 2
* Each patient must sign a study-specific informed consent form

Exclusion Criteria:

Laboratory values of:

* Platelet count <30,000/uL
* AST or ALT >2 x the upper limit of normal (ULN)
* Total bilirubin >2 x ULN
* Creatinine >2.0 mg/dL
* Chemotherapy, radiation therapy, immunotherapy, systemic corticosteroids, or systemic biologic anticancer therapy within 21 days before beginning study treatment
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States